CLINICAL TRIAL: NCT01151410
Title: A Multicenter, Double-blind, Randomized, 52-week, Extension Study to Evaluate the Long Term Safety, Tolerability and Efficacy of Aliskiren Compared to Enalapril in Pediatric Hypertensive Patients 6-17 Years of Age
Brief Title: An Extension Study to Evaluate the Long Term Safety, Tolerability and Efficacy of Aliskiren Compared to Enalapril in Pediatric Hypertensive Patients 6-17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2365E1; 2009-017029-20 (EudraCT Number)
Record Dates: First submitted 2010-06-23; First posted 2010-06-28 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
Keywords: Pediatric hypertension; primary hypertension; secondary; hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension; Neoplasm Metastasis | interventions — aliskiren; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aliskiren (Experimental): Patients will receive one of the following doses based on the their weight: Low weight (≥20 to <50 kg) patients: Starting dose 37.5 mg with optional titration to 75 and then 150 mg Mid weight (≥50 to <80 kg) patients: Starting dose 75 mg with optional titration to 150 and then 300 mg High weight (≥80 to ≤150 kg) patients: Starting dose 150 mg with optional titration to 300 and then 600 mg
  Interventions: Drug: Aliskiren
- Enalapril (Active Comparator): Patients will receive one of the following doses based on their weight: Low weight (≥20 to <50 kg) patients: Starting dose 2.5 mg with optional titration to 5 and then 10 mg Mid weight (≥50 to <80 kg) patients: Starting dose 5 mg with optional titration to 10 and then 20 mg High weight (≥80 to ≤150 kg) patients: Starting dose 10 mg with optional titration to 20 and then 40 mg
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Aliskiren — Low weight patients: Starting dose 37.5 mg with optional titration to 75 and then 150 mg
  Mid weight patients: Starting dose 75 mg with optional titration to 150 and then 300 mg
  High weight patients: Starting dose 150 mg with optional titration to 300 and then 600 mg
  Arms: Aliskiren
Drug: Enalapril — Low weight patients: Starting dose 2.5 mg with optional titration to 5 and then 10 mg
  Mid weight patients: Starting dose 5 mg with optional titration to 10 and then 20 mg
  High weight patients: Starting dose 10 mg with optional titration to 20 and then 40 mg
  Arms: Enalapril

SUMMARY:
The purpose of this study is to evaluate in a randomized, double-blind fashion, the long-term safety, tolerability and efficacy profile of aliskiren compared to the active comparator enalapril in children, 6 - 17 years old with hypertension (msSBP ≥ 95th percentile for age, gender and height, at baseline in study CSPP100A2365). Patients will be randomized to receive either aliskiren or enalapril. Weight-group based doses of aliskiren or enalapril will be administered once daily and children will receive study medication in a double-blind manner. This study is being conducted to support monotherapy registration of aliskiren for the treatment of hypertension in pediatric patients 6-17 years of age (age at baseline in Study CSPP100A2365).

ELIGIBILITY:
Inclusion Criteria:

* msSBP (mean of 3 systolic blood pressure measurements) must be ≥ 95th percentile for age, gender and height, at Visit 2 (randomization), in study CSPP100A2365
* Must be ≥ 20 kg and ≤ 150 kg at Visit 2 (randomization), in study CSPP100A2365
* Must be able to swallow minitablets (2mm in diameter) administered in soft food
* Successful completion of Phase 1 (dose response phase) and at least 1 week of Phase 2 (placebo withdrawal phase) of the CSPP100A2365 protocol, with no serious drug-related adverse event(s).

Exclusion Criteria:

* Patient receiving immunosuppressant medication (e.g. cyclosporine, MMF, etc) other than oral/topical steroids, for any medical condition
* Current diagnosis of heart failure (NYHA Class II-IV) or history of cardiomyopathy or obstructive valvular disease
* msSBP ≥ 25% above the 95th percentile
* Second or third degree heart block without a pacemaker
* AST/SGOT or ALT/SGPT >3 times the upper limit of the reference range
* Total bilirubin > 2 times the upper limit of the reference range
* Creatinine clearance < 30 mL/min/1.73m² (calculated using Modified Schwartz formula to estimate glomerular filtration rate [GFR]), based on the serum creatinine concentration obtained at the screening visit)
* WBC count < 3000/mm³
* Platelet count < 100,000/mm³
* Serum potassium > 5.2 mEq/L
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (16):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Dalton, Georgia
  - Novartis Investigative Site, Lewiston, Idaho
  - Novartis Investigative Site, Park Ridge, Illinois
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Hattiesburg, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Charleston, West Virginia
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Hungary (6):
  - Novartis Investigative Site, Nyíregyháza, Hungary
  - Novartis Investigative Site, Szeged, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, San Juan, Puerto Rico
- Slovakia (5):
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Myjava, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Trnava, Slovakia
- Novartis Investigative Site, Ankara, Turkey, Turkey (Türkiye)

REFERENCES:
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren | Enalapril
Started | 104 | 104
Safety Set (SAF) | 105 | 103 (Number of patients in SAF differed due to kit dispensing error in 1 patient at Visit 12)
Completed | 93 | 89
Not Completed | 11 | 15
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Lost to Follow-up | 3 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Protocol deviation | 2 | 1
Not completed — Administrative problems | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 1
Not completed — Abnormal laboratory value(s) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Enalapril | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (3.40) | 11.9 (3.40) | 11.8 (3.39)
Age, Customized [Number; unit: participants]
  Children 6 - 11 years | 50 | 51 | 101
  Adolescents 12 - 17 years | 54 | 53 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 32 | 72
  Male | 64 | 72 | 136

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) at to End of Study
Description: Sitting blood pressure was measured using a calibrated standard sphygmomanometer after the participants remained in sitting position for 5 minutes at clinic during the visit. The repeat sitting measurements were made at 2 to 3 minute intervals and the mean of three sSBP measurements were used as the average sitting office blood pressure for that visit.
Time Frame: Baseline - end of study (Week 52 or Last observation carried forward (LOCF)
Population: Full analysis set (FAS) included all randomized patients for this trial
Measure: Least Squares Mean (Standard Error); unit: millimeter(s) of mercury (mmHg)
Arm/Group | Aliskiren | Enalapril
Number analyzed (Participants) | 104 | 104
millimeter(s) of mercury (mmHg) | -7.63 (1.16) | -7.94 (1.14)
Statistical Analysis 1: Comparison: Aliskiren vs Enalapril; Test type: Non-Inferiority or Equivalence — Indicates statistical significance at 0.025 level for one sided non-inferiority testing at 4mmHg margin; p = 0.0040, ANCOVA; Mean Difference (Net) = 0.31, 95% CI 1-sided [lower limit -2.40]

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study
Description: Sitting blood pressure was measured using a calibrated standard sphygmomanometer after the participants remained in sitting position for 5 minutes at clinic during the visit. The repeat sitting measurements were made at 2 to 3 minute intervals and the mean of three sDBP measurements were used as the average sitting office blood pressure for that visit.
Time Frame: Baseline - end of study (Week 52 or Last observation carried forward (LOCF)
Population: Full analysis set (FAS) included all randomized patients for this trial
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren | Enalapril
Number analyzed (Participants) | 104 | 104
mmHg | -3.90 (0.87) | -4.94 (0.85)

3. Secondary Outcome: Change in Mean Arterial Pressure (MAP) (mmHg) From Baseline to End of Study
Description: MAP was defined as the average arterial pressure during a single cardiac cycle. The MAP was measured as sum of diastolic blood pressure (DBP) and one third of difference between systolic blood pressure (SBP) and DBP i.e. MAP = DBP+1/3*(SBP--DBP).
Time Frame: Baseline to end of study (Week 52 or LOCF)
Population: Full analysis set (FAS) included all randomized patients for this trial
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren | Enalapril
Number analyzed (Participants) | 104 | 104
mmHg | -5.15 (0.89) | -5.95 (0.87)

ADVERSE EVENTS:
Arm/Group | Aliskiren | Enalapril
Serious Adverse Events (participants affected / at risk) | 3/105 | 12/103
Other Adverse Events (participants affected / at risk) | 52/105 | 51/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=105) | Enalapril (N=103)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Device malfunction (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Tetany (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Psychosomatic disease (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=105) | Enalapril (N=103)
Vomiting (Gastrointestinal disorders) | 8 | 5
Pyrexia (General disorders) | 6 | 5
Bronchitis (Infections and infestations) | 5 | 7
Nasopharyngitis (Infections and infestations) | 8 | 6
Pharyngitis (Infections and infestations) | 7 | 2
Upper respiratory tract infection (Infections and infestations) | 15 | 15
Viral infection (Infections and infestations) | 10 | 8
Headache (Nervous system disorders) | 7 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single- site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.